CLINICAL TRIAL: NCT01777646
Title: A Phase IIa, Open Label, Dose-escalating Clinical Study to Evaluate the Safety, Tolerability and Therapeutic Effects of Transplantation of Autologous Mesenchymal Bone Marrow Stromal Cells Secreting Neurotrophic Factors (MSC-NTF), in Patients With Amyotrophic Lateral Sclerosis (ALS).
Brief Title: Autologous Mesenchymal Bone Marrow Stromal Cells Secreting Neurotrophic Factors (MSC-NTF), in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brainstorm-Cell Therapeutics (Industry)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-NTF-002-HMO-CTIL
Record Dates: First submitted 2012-12-12; First posted 2013-01-29 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Mesenchymal Strmal Cells (MSC); Amyotrophic Lateral Sclerosis (ALS); Neuroprotection; Neurodegeneration; Stem cells
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Nerve Degeneration

ARMS (1):
- MSC-NTF (Experimental)
  Interventions: Biological: MSC_NTF cells transplantation by multiple intramuscular injections at 24 separate sites, in addition to a single intrathechal injection into the CSF

INTERVENTIONS:
Biological: MSC_NTF cells transplantation by multiple intramuscular injections at 24 separate sites, in addition to a single intrathechal injection into the CSF

SUMMARY:
The study will evaluate the safety, tolerability and therapeutic effects of transplantation of escalating doses of autologous cultured mesenchymal bone marrow stromal cells secreting neurotrophic factors (MSC-NTF), in patients with amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
This is a phase IIa prospective, open label, dose-escalating, three patient-group clinical study, to evaluate the safety, tolerability and preliminary efficacy of autologous cultured mesenchymal bone marrow stromal cells secreting neurotrophic factors (MSC-NTF), as a potent treatment for patients with Amyotrophic Lateral Sclerosis (ALS) at the early disease stages. This study is a single center trial. It is anticipated that the study will be conducted at the Department of Neurology & Laboratory of Neuroimmunology, at the Hadassah Hebrew University Medical Center, Jerusalem in Israel. In addition, ALS patients could also be referred to the clinical site above by other medical centers.

All patients enrolled will have a documented history of ALS disease prior to study enrollment. Patients diagnosed as early stage ALS disease with duration of less than 2 years. ALS patients identified as "predisposed" will be approached and requested to sign an Informed Consent Form (ICF). Overall, 14 patients will be recruited.

Treatment will start with the lowest dose (94x106 cells) and the dose will be increased to the next medium and high dose (141x106 and 188x106 respectively), for the next patients group only following safety analysis.

The expected duration of patient screening period prior to enrollment into this study is in-between two weeks up to 2 days prior to the study enrollment day during visit 2 (verification of compliance with inclusion/exclusion criteria including clinical laboratory results). Eligible patients will be enrolled into the study and will be observed for every month during a "run in period" of 3 months for determination of the progression rate of the disease (allowing a time window of ± 5 days for all visits). During the "run in period" after about 6 weeks following enrollment, patients of both study groups will undergo a Bone Marrow Aspiration (BMA) procedure and MSC-NTF cells will be produced from the bone marrow aspirate based on Brainstorm Cell Therapeutics Ltd proprietary method. On the last "run in period" visit, patients will undergo the treatment and MSC-NTF will be transplanted by IM+IT to the early ALS patients.

After the MSC-NTF transplantation patients will be observed on a monthly basis for a post treatment follow up period of 6 months (allowing a time window of ± 5 days for all visits). Treatment safety, adverse events and exploratory parameters, to establish ALS progression rate assessment of the disease will be recorded throughout the duration of the "run in period" and the post treatment follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must fulfill El Escorial criteria (APPENDIX 2) for definite or probable ALS (sporadic and not familial)
2. Participants, either men or non pregnant women are between 20 and 75 years of age.
3. The patient is mentally intact and psychologically stable
4. Patients will be with an ALS-FRS-R scale (APPENDIX 3) of at least 30 and disease duration of less than 2 years.
5. Patient has sufficiently bulky muscles.
6. Participant understands the nature of the procedure and provides written informed consent prior to any study procedure.

Exclusion Criteria:

1. Patient has a positive test for HBV, HCV or HIV.
2. Patient has high protein in the CSF (Protein > 70 mg/ml).
3. Patient has lymphocytosis in the CSF (lymphocytes > 5/ml).
4. Patient is positive for anti-GM1 antibodies.
5. Patient has significant conduction blocks or slow nerve conduction velocities (a reduction of more than 30%) confirmed by nerve conduction velocity - EMG studies.
6. The patient is a respiratory dependent patient.
7. Patients with renal failure (Cr > 2 mg/dl).
8. Patients with impaired hepatic function (ALT, AST or GGT 2-fold higher than normal upper limit).
9. Patients suffering from significant cardiac disease, malignant disease or any other disease that may risk the patient or interfere with the ability to interpret the results
10. Patient with active infections.
11. Participation in another clinical trial within 1 month prior to start of this study.
12. Patient has not been treated previously with any cellular therapy.
13. Subject unwilling or unable to comply with the requirements of the protocol.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety evaluation and tolerability of a single treatment administration in an escalating-dose of autologous cultured mesenchymal bone marrow stromal cells secreting neurotrophic factors (MSC-NTF) | At baseline and up to 6 month following treatment administration

SECONDARY OUTCOMES:
Changes in the progression rate of the disease as evidenced by changes in the ALS functional rating scale | At baseline and up to 6 month following treatment administration
Changes in muscle strength grading (MVIC) by muscle chart | At baseline and up to 6 month following treatment administration
Changes in muscle bulk estimated by MRI of the upper and lower extremities | At baseline and up to 6 month following treatment administration
Change in upper and lower extremities circumference (cm) | At baseline and up to 6 month following treatment administration
Changes in EMG parameters | At baseline and up to 6 month following treatment administration

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Karusis, MD, PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Gothelf Y, Kaspi H, Abramov N, Aricha R. miRNA profiling of NurOwn(R): mesenchymal stem cells secreting neurotrophic factors. Stem Cell Res Ther. 2017 Nov 7;8(1):249. doi: 10.1186/s13287-017-0692-1. PMID 29116031
- [Derived] Petrou P, Gothelf Y, Argov Z, Gotkine M, Levy YS, Kassis I, Vaknin-Dembinsky A, Ben-Hur T, Offen D, Abramsky O, Melamed E, Karussis D. Safety and Clinical Effects of Mesenchymal Stem Cells Secreting Neurotrophic Factor Transplantation in Patients With Amyotrophic Lateral Sclerosis: Results of Phase 1/2 and 2a Clinical Trials. JAMA Neurol. 2016 Mar;73(3):337-44. doi: 10.1001/jamaneurol.2015.4321. PMID 26751635